CLINICAL TRIAL: NCT02853084
Title: An Open Label, Single Arm Trial to Evaluate the Efficacy, Safety, and Pharmacokinetics of HL2351 in Patients With Cryopyrin Associated Periodic Syndromes
Brief Title: HL2351 CAPS Phase II Study
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: difficult of recruiting
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HL_C201
Record Dates: First submitted 2016-05-10; First posted 2016-08-02 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-05

CONDITIONS: Cryopyrin-Associated Periodic Syndromes (CAPS)
Keywords: Auto-inflammatory diseases; IL-1 inhibitors; HL2351; Cryopyrin-Associated Periodic Syndromes (CAPS); Neonatal Onset Multisystem Inflammatory Disease (NOMID); Muckle-Wells Syndrome (MWS); Familial Cold Autoinflammatory Syndrome (FCAS)
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HL2351 (Experimental)
  Interventions: Drug: HL2351

INTERVENTIONS:
Drug: HL2351 — The dose will be adjusted based on disease activities

SUMMARY:
This is an open label, single arm trial to evaluate the efficacy, safety, and pharmacokinetics of HL2351 in patients with cryopyrin associated periodic syndromes (CAPS).

DETAILED DESCRIPTION:
This trial enrolls patients with CAPS being on stable dose of anakinra daily and then switch over HL2351 given once weekly. It consists of 4 phases, 6-week screening, single dose PK, 6-month multiple dose, and 18-month extension phase.

ELIGIBILITY:
Inclusion Criteria:

* Documented molecular diagnosis of NALP3 mutation or diagnosis of CAPS based on sign and symptom
* Diagnosis of CAPS based on signs and symptoms
* Current stable doses of anakinra, alone or in combination with methotrexate or corticosteroids

Exclusion Criteria:

* Patient been diagnosed with a hereditary periodic fever syndrome or autoinflammatory disease other than CAPS
* Patients whose disease is inadequately controlled on current stable doses of anakinra, alone or in combination with methotrexate or corticosteroids

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2015-10; Primary Completion 2017-05 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Change in Diary Symptom Sum Score (DSSS) | from baseline to Month 6
Change in SAA, CRP, ESR levels | from baseline to Month 6, from baseline to each visit up to Month 24
Change in physician's global assessment of autoinflammatory using 100mm VAS score disease | from baseline to Month 6, from baseline to each visit up to Month 24
Change in patient's(parents or legal guardians) global assessment of autoinflammatory using 100mm VAS score disease | from baseline to Month 6, from baseline to each visit up to Month 24
Pharmacokinetic profile(Cmax) | 0,12,24,36,48,72,96,144,168 hr
Pharmacokinetic profile(AUClast) | 0,12,24,36,48,72,96,144,168 hr
Pharmacokinetic profile(AUCinf) | 0,12,24,36,48,72,96,144,168 hr
Pharmacokinetic profile(Tmax) | 0,12,24,36,48,72,96,144,168 hr
Pharmacokinetic profile(t1/2) | 0,12,24,36,48,72,96,144,168 hr

CONTACTS AND LOCATIONS:
Overall Officials: JOONG GON KIM, Principal Investigator — Seoul National University Hospital
Locations (1):
- Handok Inc., Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided